CLINICAL TRIAL: NCT01128413
Title: Emergency Department (ED) Flow-directed Fluid Optimization Resuscitation Trial (EFFORT)
Acronym: EFFORT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Christopher Holthaus, MD, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFFORT-10-0593
Record Dates: First submitted 2010-05-06; First posted 2010-05-21 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Shock
Keywords: Shock; Resuscitation; Hemodynamics; Emergencies; Critical Care; Lactic Acid; Plasma volume
MeSH Terms: conditions — Shock; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluid Optimization (FO) (Experimental): Cheetah NICOM® (non-invasive cardiac output monitoring) Passive Leg Raise Testing (PLRT) that demonstrates a >/= 15% change in stroke volume index (SVI) or cardiac index (CI) will receive a 500ml normal saline bolus. NICOM® PLRT with SVI or CI <15% will receive a saline lock. If bolused, NICOM® PLRT will be performed within 10 minutes after the bolus with the decision to re-bolus or saline lock according to repeated NICOM® PLRT measurements. If saline locked, NICOM® PLRT will be performed every 30 minutes with the decision to re-bolus or saline lock according to repeated NICOM® PLRT measurements.
  Additionally, USCOM®, IVC Ultrasound collapsibility, CURVES Questionnaire, and repeat lactate measurements will be performed.
  Interventions: Device: Cheetah NICOM® PLRT; Device: USCOM ® (Ultrasound Cardiac Output Monitor); Device: Inferior Vena Cava (IVC) Ultrasound Collapsibility; Behavioral: CURVES Questionnaire; Biological: Lactate Clearance; Biological: 500ml Normal Saline Bolus
- Routine Care (RC) (Active Comparator): Patients randomized to receive routine ED care will receive IV fluid administration per the treating clinicians discretion. The Cheetah NICOM®PLRT, USCOM®, IVC Ultrasound collapsibility, and CURVES Questionnaire will be performed and repeat lactate measurements will only be revealed to the routine care arm if they are used as part of the provider's routine care.
  Interventions: Device: Cheetah NICOM® PLRT; Device: USCOM ® (Ultrasound Cardiac Output Monitor); Device: Inferior Vena Cava (IVC) Ultrasound Collapsibility; Behavioral: CURVES Questionnaire; Biological: Lactate Clearance; Biological: Clinician Discretion Intravenous Fluid Management

INTERVENTIONS:
Device: Cheetah NICOM® PLRT — Cheetah NICOM® (non-invasive cardiac output monitoring)PLRT (passive leg raise testing) protocol: The patient while in a semi-recumbent position (legs level, torso up 45 degrees) will have 3 minutes of stroke volume and cardiac index monitoring. Following the 3 minutes, the patient will be placed in a leg raised position (torso level, legs up 45 degrees) for 3 minutes of stroke volume and cardiac index monitoring. NICOM® PLRT will be performed within 10 minutes after any fluid bolus in both arms with results blinded to the Routine Care arm. If saline locked or maintenance IV fluid rate, NICOM® PLRT will be performed every 30 minutes in both arms with results blinded to the Routine Care arm.
Device: USCOM ® (Ultrasound Cardiac Output Monitor) — Patients while in the Cheetah NICOM® PLRT semi-recumbent position (legs level, torso up 45 degrees) will have simultaneous USCOM® stroke volume and cardiac index monitoring. Following the 3 minutes of Cheetah NICOM® PLRT semi-recumbent positioning, the patient will be placed in a leg raised position (torso level, legs up 45 degrees) and have simultaneous USCOM® stroke volume and cardiac index monitoring. USCOM® monitoring will be blinded to the Routine Care arm unless used as part of a provider's routine practice. USCOM® changes in SVI or CI with PLRT will be calculated after the patient leaves the ED.
Device: Inferior Vena Cava (IVC) Ultrasound Collapsibility — Patients while in the Cheetah NICOM® PLRT semi-recumbent position (legs level, torso up 45 degrees) will have a simultaneous 6-12 second ultrasound recording of their IVC. These recordings will be reviewed later by an ultrasonographer and graded for volume responsiveness. The reviewing ultrasonographer will be blinded to the Cheetah NICOM® PLRT results.
Behavioral: CURVES Questionnaire — The CURVES (CardiovascUlar Response & Volume Estimation in Shock) Questionnaire consists of multiple provider questions aimed at defining the presumed shock etiology and anticipated responses to interventions. This will be administered to both arms.
Biological: Lactate Clearance — Lactate samples will be drawn at time 0, 1, 3, & 6 hours (or at ED departure if before 6 hours). Time 0 lactate will be revealed to the Routine Care arm and subsequent lactates revealed to the Routine Care arm only if serial lactates are part of the provider's routine practice.
Biological: 500ml Normal Saline Bolus — Patients randomized to the experimental arm and having a >/= 15% change in stroke volume index (SVI) or cardiac index (CI) via Cheetah NICOM®PLRT will be given a 500ml normal saline fluid bolus.
  Arms: Fluid Optimization (FO)
Biological: Clinician Discretion Intravenous Fluid Management — Clinicians caring for patients randomized to the Routine Care arm will within 10 minutes after any fluid bolus be asked to decide via their clinical discretion if they want to re-bolus, saline lock, or place the patient on a maintenance IV fluid rate. If the patient is on a saline lock or maintenance fluid rate, clinicians will be asked every 30 minutes to decide via their clinical discretion to re-bolus, saline lock, or place the patient on a maintenance IV fluid rate.
  Arms: Routine Care (RC)

SUMMARY:
The short term goal of this study is to evaluate a non-invasive approach that optimizes intravenous (IV) fluid administration according to heart performance and results in surrogate improvements in morbidity and mortality via lactate clearance. Additional objectives include comparative assessments of methods for determining volume responsiveness and establishing a prevalence of volume responsive shock in the Emergency Department (ED).

DETAILED DESCRIPTION:
Patients will be randomized to Routine Care (RC) or Fluid Optimizations (FO) arms. Both arms will have interval Cheetah NICOM® (non-invasive cardiac output monitoring) Passive Leg Raise Testing (PLRT).

In the FO arm, patients having a PLRT demonstrating a >/= 15% change in stroke volume index (SVI) or cardiac index (CI) patients will receive a 500ml normal saline bolus. If the NICOM® PLRT shows a SVI or CI <15% patients will receive a saline lock. If bolused, NICOM® PLRT will be performed within 10 minutes after the bolus with the decision to re-bolus or saline lock according to repeated NICOM® PLRT measurements. If saline locked, NICOM® PLRT will be performed every 30 minutes with the decision to re-bolus or saline lock according to repeated NICOM® PLRT measurements.

In the RC arm, IV fluid administration will be per the treating clinicians discretion. The Cheetah NICOM®PLRT will be performed before and after each clinician fluid bolus.

Lactate blood samples will be drawn at time zero, 1 hour, 3 hours, 6 hours, and/or ED departure and compared between arms.

ELIGIBILITY:
Inclusion Criteria:

* Hypotension (Systolic Blood Pressure ≤90mm Hg or Mean Arterial Pressure ≤ 65 mm Hg) after ≥ 20ml/kg fluids OR
* Vasopressor Use OR
* Lactate ≥ 2.5 mmol/L

Exclusion Criteria:

* Pulse Oximetry <90% despite supplemental oxygen or intubation
* Seizure in the last 24 hours
* Prisoner
* Pregnancy
* Age <18
* Allergy to coupling or ultrasound gel
* Inability to do passive leg raise
* Inability to obtain IV access
* Treating clinician discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher V Holthaus, MD, Principal Investigator — Washington University School of Medicine; Brian M Fuller, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital Emergency Department, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinert R, Spektor M. Evidence-based emergency medicine/rational clinical examination abstract. Clinical assessment of hypovolemia. Ann Emerg Med. 2005 Mar;45(3):327-9. doi: 10.1016/j.annemergmed.2004.09.021. No abstract available. PMID 15726060
- [Background] Jones AE, Kline JA. Use of goal-directed therapy for severe sepsis and septic shock in academic emergency departments. Crit Care Med. 2005 Aug;33(8):1888-9; author reply 1889-90. doi: 10.1097/01.ccm.0000166872.78449.b1. No abstract available. PMID 16096485
- [Background] Blow O, Magliore L, Claridge JA, Butler K, Young JS. The golden hour and the silver day: detection and correction of occult hypoperfusion within 24 hours improves outcome from major trauma. J Trauma. 1999 Nov;47(5):964-9. doi: 10.1097/00005373-199911000-00028. PMID 10568731
- [Background] Shapiro NI, Howell MD, Talmor D, Nathanson LA, Lisbon A, Wolfe RE, Weiss JW. Serum lactate as a predictor of mortality in emergency department patients with infection. Ann Emerg Med. 2005 May;45(5):524-8. doi: 10.1016/j.annemergmed.2004.12.006. PMID 15855951
- [Background] Nguyen HB, Rivers EP, Knoblich BP, Jacobsen G, Muzzin A, Ressler JA, Tomlanovich MC. Early lactate clearance is associated with improved outcome in severe sepsis and septic shock. Crit Care Med. 2004 Aug;32(8):1637-42. doi: 10.1097/01.ccm.0000132904.35713.a7. PMID 15286537
- [Background] Jones AE, Shapiro NI, Trzeciak S, Arnold RC, Claremont HA, Kline JA; Emergency Medicine Shock Research Network (EMShockNet) Investigators. Lactate clearance vs central venous oxygen saturation as goals of early sepsis therapy: a randomized clinical trial. JAMA. 2010 Feb 24;303(8):739-46. doi: 10.1001/jama.2010.158. PMID 20179283
- [Background] Sinclair S, James S, Singer M. Intraoperative intravascular volume optimisation and length of hospital stay after repair of proximal femoral fracture: randomised controlled trial. BMJ. 1997 Oct 11;315(7113):909-12. doi: 10.1136/bmj.315.7113.909. PMID 9361539
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008 Jul;134(1):172-8. doi: 10.1378/chest.07-2331. PMID 18628220
- [Background] Marik PE, Cavallazzi R, Vasu T, Hirani A. Dynamic changes in arterial waveform derived variables and fluid responsiveness in mechanically ventilated patients: a systematic review of the literature. Crit Care Med. 2009 Sep;37(9):2642-7. doi: 10.1097/CCM.0b013e3181a590da. PMID 19602972
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429
- [Background] Thiel SW, Kollef MH, Isakow W. Non-invasive stroke volume measurement and passive leg raising predict volume responsiveness in medical ICU patients: an observational cohort study. Crit Care. 2009;13(4):R111. doi: 10.1186/cc7955. Epub 2009 Jul 8. PMID 19586543
- [Background] Corley A, Barnett AG, Mullany D, Fraser JF. Nurse-determined assessment of cardiac output. Comparing a non-invasive cardiac output device and pulmonary artery catheter: a prospective observational study. Int J Nurs Stud. 2009 Oct;46(10):1291-7. doi: 10.1016/j.ijnurstu.2009.03.013. Epub 2009 May 6. PMID 19423107
- [Background] Nguyen HB, Losey T, Rasmussen J, Oliver R, Guptill M, Wittlake WA, Corbett SW. Interrater reliability of cardiac output measurements by transcutaneous Doppler ultrasound: implications for noninvasive hemodynamic monitoring in the ED. Am J Emerg Med. 2006 Nov;24(7):828-35. doi: 10.1016/j.ajem.2006.05.012. PMID 17098106
- [Background] Barbier C, Loubieres Y, Schmit C, Hayon J, Ricome JL, Jardin F, Vieillard-Baron A. Respiratory changes in inferior vena cava diameter are helpful in predicting fluid responsiveness in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1740-6. doi: 10.1007/s00134-004-2259-8. Epub 2004 Mar 18. PMID 15034650
- [Background] Feissel M, Michard F, Faller JP, Teboul JL. The respiratory variation in inferior vena cava diameter as a guide to fluid therapy. Intensive Care Med. 2004 Sep;30(9):1834-7. doi: 10.1007/s00134-004-2233-5. Epub 2004 Mar 25. PMID 15045170
- [Background] Perera P, Mailhot T, Riley D, Mandavia D. The RUSH exam: Rapid Ultrasound in SHock in the evaluation of the critically lll. Emerg Med Clin North Am. 2010 Feb;28(1):29-56, vii. doi: 10.1016/j.emc.2009.09.010. PMID 19945597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients screened and study performed in the ED from July 2010 to November 2013.
Groups:
- Fluid Optimization (FO): Cheetah NICOM® (non-invasive cardiac output monitoring) Passive Leg Raise Testing (PLRT) that demonstrates a >/= 15% change in stroke volume index (SVI) or cardiac index (CI) will receive a 500ml normal saline bolus. NICOM® PLRT with SVI or CI <15% will receive a saline lock.
- Routine Care (RC): Patients randomized to receive routine ED care. IV fluid administration will be per the treating clinicians discretion.
Period: Overall Study
Arm/Group | Fluid Optimization (FO) | Routine Care (RC)
Started | 11 | 11
Completed | 7 | 10
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — NICOM Monitor Problems | 2 | 1
Not completed — Pt made DNR | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Optimization (FO) | Routine Care (RC) | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 4 | 4 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [47 to 66] | 59 [54 to 65] | 57 [51 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Lactate Clearance
Description: The median lactate clearance from time zero to within 6 hours of the ED stay.
Time Frame: The median lactate clearance within 6 hours of the ED stay.
Population: Only 9 total patients (5 Fluid Optimization; 4 Routine Care) stayed in the Emergency Department for a full 6 hours to allow calculation of a 6 hour lactate clearance. The rest of the patients left were dispositioned out of the ED before the 6 hour mark and therefore unable to calculate a 6 hour lactate clearance.
Measure: Median (Inter-Quartile Range); unit: percent lactate clearance
Arm/Group | Fluid Optimization (FO) | Routine Care (RC)
Number analyzed (Participants) | 5 | 4
percent lactate clearance | 54 [19 to 57] | 56 [49 to 59]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Inpatient records reviewed for death within 24 hours of study enrollment, disability, worsening oxygenation and/or escalation of monitoring and/or supportive care believed to be directly related to excess IV fluid administration, electrode adhesive or ultrasound gel hypersensitivity, IV site infection or inflammation.
Arm/Group | Fluid Optimization (FO) | Routine Care (RC)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Trial terminated early due to lack of resources leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No